CLINICAL TRIAL: NCT04194242
Title: A Phase I, Single Center, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Access the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HEC96719 Tablets in Chinese Healthy Volunteers
Brief Title: The Tolerability , Pharmacokinetics and Pharmacodynamics Study of HEC96719 Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC96719-P-01/CRC-C1931
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2019-12

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEC96719 tablets (Experimental): Including 7 dose groups(0.1、0.2、0.5、1、2、3、4 mg).Each dose group was given only once.After an overnight stay of at least 10h on an empty stomach, 240 mL of water was administered in the morning under the condition of an empty stomach. Water was forbidden for 1h before and 1h after administration, and fasting for 4h after administration.
  Interventions: Drug: HEC96719 tablets
- placebo tablets (Placebo Comparator): Including 7 dose groups(0.1、0.2、0.5、1、2、3、4 mg).Each dose group was given only once.After an overnight stay of at least 10h on an empty stomach, 240mL of water was administered in the morning under the condition of an empty stomach. Water was forbidden for 1h before and 1h after administration, and fasting for 4h after administration.
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: HEC96719 tablets — 0.1、0.2、0.5、1、2、3、4 mg HEC96719 tablet in day1
  Arms: HEC96719 tablets
Drug: Placebo tablet — 0.1、0.2、0.5、1、2、3、4 mg Placebo tablet in day1
  Arms: placebo tablets

SUMMARY:
This study is a safety, tolerability, and pharmacokinetics phase Ⅰstudy of HEC96719, in healthy subjects.This study is the healthy adult subjects single ascending-dose research

DETAILED DESCRIPTION:
This study will evaluate the safety and tolerability of escalating single oral doses of HEC96719, and characterize the single-dose pharmacokinetics (PK) of HEC96719. Participants will receive either HEC96719 or HEC96719 placebo.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study, able to understand and sign the informed consent, and able to complete the the study in accordance with the requirements of the study.
* Female subjects who are not pregnant or lactating and male subjects whose female partners are fertile shall voluntarily take effective contraceptive measures from the date of signing the informed consent form to 3 months after the medication.
* When signing the informed consent, 18 years old ≤the age≤45 years old(including the critical value), gender is not limited.
* Male body weight ≥50kg, female body weight ≥45kg, and body mass index (BMI) in the range of 18-28 kg/m2 (including the critical value).
* No clinical significance of vital signs, physical examination, laboratory examination, electrocardiogram, ultrasound abdomen and chest X-ray (posterior and anterior) results.

Exclusion Criteria:

* Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis.
* Those who are known to have allergy history or allergy constitution to the test preparation and any of its components or related preparations.
* Intemperant or regular drinkers within 3 months prior to the study, i.e., those who consumed more than 21 units of alcohol per week (1 unit =360mL beer or 45mL spirit with 40% alcohol or 150mL wine), or those who were positive on the alcohol breath test.
* Those who had a blood donation or blood loss of >400mL within one month before taking the study drug.
* Those who have participated in clinical trials of other drugs within 3 months before randomization.
* Subjects considered by the investigator to have other factors unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Adverse events of the single ascending-dose | From the baseline to day7
  To assess the safe and tolerability of the single ascending-dose

SECONDARY OUTCOMES:
Cmax | At pre-defined intervals from Days 1-2
  Maximum Plasma Concentration(Cmax)of HEC96719 in single ascending dose
AUC | At pre-defined intervals from Days 1-2
  Area Under the Curve(AUC) of HEC96719 in single ascending dose
Tmax | At pre-defined intervals from Days 1-2
  Maximum Peak Time(Tmax) of HEC96719 in single ascending dose
T1/2 | At pre-defined intervals from Days 1-2
  Terminal elimination half-life(T1/2) of HEC96719 in single ascending dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Shanghai xuhui district central hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No